CLINICAL TRIAL: NCT03713190
Title: A Phase II,Randomized,Cross-over,Double-blind, Placebo- Controlled,Single Center Study of the Effect of Empagliflozin a SGLT-2 Inhibitor,on Endogenous Glucose Production and Plasma Glucagon Levels in Patients With ESRD
Brief Title: Effects of Empagliflozin on Endogenous Glucose Production in End Stage Renal Disease(ESRD).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Prof. Stefano Del Prato, Clinical Resercher, University of Pisa
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EMPA-1
Record Dates: First submitted 2018-07-18; First posted 2018-10-19 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Active Comparator): SGLT-2 inhibitor
  Interventions: Combination Product: Empagliflozin
- placebo (Placebo Comparator): A substance without specific pharmacology principles.
  Interventions: Combination Product: Empagliflozin; Drug: Placebo

INTERVENTIONS:
Combination Product: Empagliflozin — Sodium-glucose co-transporter 2 (SGLT2), a low-affinity, high-capacity member of an increasingly numerous family of co-transporters, is highly expressed in the proximal renal tubule, and account for the majority of the reabsorption of filtered glucose.
Drug: Placebo — A substance without specific pharmacology principles
  Arms: placebo

SUMMARY:
A study of the effects of empagliflozin, a SGLT-2 inhibitor, on endogenous glucose production and plasma glucagon levels in patients with end-stage renal disease (ESRD)

DETAILED DESCRIPTION:
The impact of SGLT-2 inhibition on endogenous glucose production and plasma glucagon levels will be compared measured in patients with ESRD.The secondary endpoints are the mean difference in plasma glucose, insulin, c-peptide, FFA,GH, epinephrine, norepinephrine, cortisol and blood pressure during the last hour of the experiment between empagliflozin versus placebo administration in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Age = 30-70 years
3. BMI< 40 Kg/m 2 and stable weight (± 3 lbs) over the preceding three months
4. Normal Glucose Tolerance (HbA1c > 4.5 % and < 5.7%) or Type 2 diabetes (HbA1c >5.7 % and <10.0%)
5. End Stage Renal Disease (GFR <15 ml/min/1.73 m 2 or hemodialysis)
6. Subjects are capable of giving informed consent

Exclusion Criteria:

1. Prednisone treatment
2. Beta blocker or any medication that affects sympathetic/parasympathetic activity
3. Known Empagliflozin Excipient Hypersensitivity
4. Liver function enzymes higher more than two times the upper limit
5. Ongoing urinary tract infection
6. history of cancer of any type;
7. cerebrovascular or symptomatic peripheral vascular disease;
8. heart disease class III or IV NYHA;
9. Type 1 Diabetes
10. drug or alcohol abuse;
11. life expectancy <3 yrs
12. blood pressure >150/100 mmHg
13. Donation of blood to a blood bank, blood transfusion, or participation in a clinical study requiring withdrawal of > 400 mL of blood during the 8 weeks prior to the enrollment visit and at least 8 weeks thereafter
14. Women of child bearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study (estrogen and/or progesterone treatment)
15. Patient with a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance which, in the opinion of the investigator or coordinator, might pose an unacceptable risk to the patient or interfere with trial procedures

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Changes in plasma Glucose level | 2 hours
  Because of their mechanism of action, SGLT-2 inhibitor efficacy to reduce plasma glucose level is highly dependent upon renal function. With GFR decreasing, glucose tubular load will decrease and less glucose will be reabsorbed because of SGLT2-inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Del prato, Principal Investigator — University of Pisa
Locations (1):
- Department of Endocrinology and Metabolism, University of Pisa, Pisa, Italy